CLINICAL TRIAL: NCT06662032
Title: Randomized Clinical Investigation to Assess Preliminary Clinical Performance, Effectiveness and Safety of the LumbaCure® (Prototype C190070.01) Medical Device When Used in Patients Suffering From Chronic Low Back Pain
Brief Title: Clinical Investigation to Assess the Clinical Effect of the LumbaCure® Intervention on Patients Suffering From Chronic Low Back Pain
Acronym: LumbaCure2302
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LumbaCure2302_2.0; CIV-23-05-043012 (Other: AFMPS)
Record Dates: First submitted 2024-10-16; First posted 2024-10-28 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: LBP; rehab; nCLPB

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Intervention (Experimental): In the intervention arm, participants will follow the standard rehabilitation programme at a frequency of ideally 2 times a week. LumbaCure® device will be used in addition to the standard programme. A session of 15 min will be performed at each rehabilitation session. The device is to be used by the Physiotherapist at the rehabilitation centre. In total, the participant should perform 26 LumbaCure® sessions during the intervention period, this corresponds to the number of rehabilitation sessions considered in the intervention period.
  Interventions: Device: LumbaCure®; Other: Rehab program
- Control Intervention (Active Comparator): Participants in the control arm will follow the standard rehabilitation programme at a frequency of ideally 2 times a week. To align with the duration of the intervention arm, participants in the control arm will also perform an additional 15 minutes of exercises (following standard care of the site).
  Interventions: Other: Rehab program

INTERVENTIONS:
Device: LumbaCure® — LumbaCure® is a robotic system that systematically moves the spine of affected patients with a complex proprietary algorithm.
  Arms: Test Intervention
Other: Rehab program — Standard rehabilitation program

SUMMARY:
Low Back Pain (LBP) is one of the common causes of morbidity worldwide, with a one-month prevalence of 23.3 %. Number of people with LBP reached 577 million people in 2020. LBP has been the leading cause of years lived with disability from 1990 to 2017. The highest incidence of LBP is in people in their third decade of age. LBP is a complex disease difficult to treat as most of these cases (80 - 90 %) are classified as non-specific meaning that the pain cannot be attributed to any specific injury or pathology.

Until now exercise therapy is commonly used as the treatment of choice in the rehab program of LBP. The aim of physical treatment is to improve function and prevent disability from getting worse.

LumbaCure® is a robotic system driven by a proprietary movement algorithm to induce a specific and controlled mobilization of the low back in patient requiring treatment by physical exercises due to orthopedic disorder, especially low back pain.

In Belgium, the standard back-school programme (rehabilitation programme) includes 35 rehabilitation sessions of 2 h delivered 2x/week at the investigator site (whom the first session is the inclusion visit, no therapy performed) and one session to tackle the psychological component of the condition (information on how to cope with pain). Participants are divided into two groups: the intervention group uses the LumbaCure® device (a seat that mobilizes the lower back for 15 minutes) in addition to the standard sessions (from session 2 to 27), while the control group follows the standard program with an extra 15 minutes of exercises. After session 27 (around 13 weeks), all participants continue their programme without the LumbaCure®, and their progress is assessed before the final 35th session.

DETAILED DESCRIPTION:
Low Back Pain (LBP) is one of the most common causes of morbidity worldwide, with a one-month prevalence of 23.3%. In 2020, the number of people suffering from LBP reached 577 million. From 1990 to 2017, LBP remained the leading cause of years lived with disability. The highest incidence of LBP is observed in individuals in their third decade of life. LBP is a complex condition that is often difficult to treat, as 80-90% of cases are classified as non-specific, meaning the pain cannot be attributed to a specific injury or pathology. Exercise therapy is currently the most common treatment for LBP rehabilitation, aiming to improve function and prevent the worsening of disability.

The study involves a standard rehabilitation program in Belgium consisting of 35 multidisciplinary sessions, each lasting 2 hours. Participants are divided into two groups: the intervention group and the control group. The intervention group follows the standard rehabilitation program but also uses the LumbaCure® device, a robotic system driven by a proprietary movement algorithm. The device is designed to induce controlled mobilization of the lower back, which is particularly beneficial for patients requiring physical treatment due to orthopedic disorders like low back pain. During each rehabilitation session, participants in the intervention group perform a 15-minute session on the LumbaCure® device under the supervision of a physiotherapist. Over the intervention period, participants in the intervention group are expected to complete 26 LumbaCure® sessions.

In the control group, participants follow the same standard rehabilitation program with a frequency of ideally twice a week. To match the duration of the intervention group's additional LumbaCure® sessions, participants in the control group perform 15 minutes of additional exercises based on the standard care practices of their respective rehabilitation center.

After session 27, which ideally take place over a period of 13 weeks, all participants continue with the remaining 8 sessions of the standard rehabilitation program. However, during this final phase, no LumbaCure® sessions are included for the intervention group. Participants' progress is monitored throughout the study, with a final evaluation taking place before the completion of the 35th session. This follow-up allows researchers to assess the overall effectiveness of the rehabilitation program, including the impact of the LumbaCure® device on patient outcomes compared to the standard care protocol.

ELIGIBILITY:
Inclusion Criteria:

* Chronic non-specific LBP (without red flag)
* LBP is the principal musculoskeletal condition
* Aged between 18 and 85 years old
* Able to read and understand questionnaires and communicate with the physiotherapist.
* Average Back Pain intensity over the last week above 2, assessed on Numerical Pain Rating Scale from 0 to 10 anchored with "no pain" at 0 and "worst pain imaginable " at 10.

Exclusion Criteria:

* Suspected or confirmed serious pathology (i.e infection, fracture, cancer, inflammatory arthritis, ….)
* Significant sciatica VAS > 7
* Radiculopathy
* Cognitive impairment that precludes participant from consenting, completing investigation questionnaires or complying with recommendations
* Previous spine surgery in the last 3 months
* Pregnant women
* body weight > 120 kg
* Neurological disease
* Fibromyalgia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Disability | Around week 13 (intervention period)
  Comparison of the Oswestry Disability Index (ODI) evolution from baseline to session 26 (visit 4, end of intervention) between the two treatment arms.

SECONDARY OUTCOMES:
Disability | Around week 4, 9 (intervention period) and week 18 (follow-up)
  - Comparison of the difference in the ODI evolution from baseline to session 8 (visit2) session 18 (visit 3) and during the follow-up period (visit 5), between the two treatment arms.
Back pain | Around week 4, 9, 13, 18
  * Changes from baseline, in average back pain intensity over the last week, assessed on Numerical Pain Rating Scale (NPRS) from 0 to 10. Assessed at the different timepoints (visits 2 to 4).
  * Changes in average back pain intensity over the last week, assessed on Numerical Rating Scale from 0 to 10, during the follow-up period (V5).
Function | Around week 4, 9, 13, 18
  * Change in function score, assessed using the Patient Specific Functional Scale, between baseline, and the different time points (visits 2 to 4). The PSFS requires participants to identify three problematic activities and to rate these activities on a scale from 0 to 10. A high score indicates a greater ability to accomplish the task.
  * Change in function score during the follow-up period, assessed using the Pain Specific Functional Scale.
Kinesiophobia | Around week 4, 9, 13, 18
  * Change in fear of movements and attitudes and behaviour towards pain score, evaluated through the Tampa questionnaire (TSK-17) between baseline to the different timepoints (visits 2 to 4). The total score is calculated by adding up 17 sub-questions assessed using a 4-point Likert scale (from 1 to 4), with high scores indicating a greater degree of kinesiophobia.
  * Change in fear of movements and attitudes and behaviour towards pain score, evaluated through the Tampa questionnaire,during the follow-up period (V5)
Pain catastrophizing | Around week 4, 9, 13, 18
  Change in pain catastrophizing score, evaluated through the Pain catastrophizing scale (PCS), between baseline to the different timepoints (visits 2 to 4 and during follow-up : V5). The total score is calculated by adding up 13 sub-questions assessed using a 5-point Likert scale (from 0 to 4), with high score indicating a greater degree of pain catastrophising.
Flexibility | Around week 4, 9, 13, 18
  The ability of the patient to flex the lower back via fingertips to floor distance.
  It will be performed at each visit for both groups.
Disability | Around week 4, 9 (intervention period) and week 18 (follow-up)
  - Disability Responding rate: Number and percentage of patients presenting a clinically significant improvement in the ODI at the different timepoints versus baseline in the two treatment arms
Back pain | Around week 4, 9, 13, 18
  - Pain responding rate : Number and percentage of patients presenting a clinically significant improvement in the NPRS at the different timepoints versus baseline in the two treatment arms
Function | Around week 4, 9, 13, 18
  Function responding rate : Number and percentage of patients presenting a clinically significant improvement in the pain specific function scale at the different timepoints versus baseline in the two treatment arms.
Kinesiophobia | Around week 4, 9, 13, 18
  Responding Rate kinesiophobia : Number and percentage of patients presenting a clinically significant improvement in Tampa scale (TSK-17) at the different timepoints versus baseline in the two treatment arms.
Pain catastrophizing | Around week 4, 9, 13, 18
  Responding Rate pain catastrophization : Number and percentage of patients presenting a clinically significant improvement in Pain catastrophizing scale (PCS) at the different timepoints versus baseline, in the two-treatment arms.

OTHER OUTCOMES:
Patient satisfaction | Around week 13
  For both arms, a single score of satisfaction will be calculated at the end of the intervention period based on a set of two questions: > How satisfied or dissatisfied are you with the ability of the programme to improve your low back pain condition (7-points scale)? Number and percentage of patients with a satisfaction score > 4 in the two treatment arms.
  Only for the intervention arm:
  > How globally would you rate your experience, on the LumbaCure® device (7-points scale)? Number and percentage of patients with a score > 4
Flexion/extension amplitudes and forces | Around week 0, 9, 13
  Flexion/extension amplitudes and forces measured using the Tergumed or DavidBack device. It will be performed at baseline (V1), mid-intervention (V3) and at the end of rehabilitation programme (V5) for both groups.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Jessa Ziekenhuis, Hasselt
  - Jessa Ziekenhuis, Herk-de-Stad

IPD SHARING:
Plan to Share IPD: No